CLINICAL TRIAL: NCT00430664
Title: A Comparative Study of the Safety and Efficacy of Face Talc Slurry and Iodopovidone for Pleurodesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7134-PG-1Tg-05/5469-71
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2007-02-02 (Estimated); Status verified 2007-02

CONDITIONS: Malignant Pleural Effusions; Recurrent Pleural Effusions; Primary Spontaneous Pneumothorax; Secondary Spontaneous Pneumothorax
Keywords: pleurodesis; talc; iodopovidone
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Effusion; Pneumothorax | interventions — Pleurodesis; Povidone-Iodine

INTERVENTIONS:
Procedure: Pleurodesis with either talc or iodopovidone

SUMMARY:
Pleurodesis is a technique used to fuse the two layers of the lining over the lung. This is done to get rid of collections of fluid or air in this space. A common reason would be cancer of the underlying lung or elsewhere causing fluid to collect in the pleural space. In this situation it is a palliative procedure to free the patient from symptoms like breathlessness.

DETAILED DESCRIPTION:
Pleurodesis is a technique used to fuse the two layers of the pleura. This is done to prevent reaccumulation of collections of fluid or air in this space. Common indications are malignant pleural effusions, recurrent pneumothorax and even benign effusions which are otherwise difficult to eradicate.

ELIGIBILITY:
Inclusion Criteria:

* Age over 12 years
* Symptomatic recurrent pleural effusion
* Pneumothorax needing pleurodesis

Exclusion Criteria:

* Life expectancy <1 month
* Unwilling to give consent
* Empyema
* ICTD drain output >150 ml/d
* Presence of an airleak

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2006-01; Study Completion 2007-12

PRIMARY OUTCOMES:
Success
Failure

SECONDARY OUTCOMES:
Death
Pain by VAS
Time to Pleurodesis
Others

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Gupta, MD, DM, FCCP, Principal Investigator — Additional Professor, Dept of Pulmonary Medicine, PGIMER, Chandigarh, India
Locations (1):
- PGIMER, Chandigarh, India